CLINICAL TRIAL: NCT02153788
Title: A Randomized, Double Blind, Placebo Controlled Study to Assess the Efficacy and Safety of Temazepam in HIV Seropositive Patients With Insomnia
Brief Title: Efficacy and Safety of Temazepam in HIV Seropositive Patients With Insomnia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00018356
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Results first posted 2015-03-10 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-01

CONDITIONS: Insomnia
Keywords: Insomnia; HIV
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Temazepam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- temazepam (Active Comparator): After screening, all subjects meeting entry criteria will be placed on the same single blind study drug treatment, asked to complete a daily sleep diary, and return one week later. After one week subjects randomized to temazepam will be given temazepam 15 mg for 12 weeks.
  Interventions: Drug: Temazepam
- Placebo (Placebo Comparator): After screening, all subjects meeting entry criteria will be placed on the same single blind study drug treatment, asked to complete a daily sleep diary, and return one week later. After one week subjects randomized to placebo will be given placebo for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Temazepam — Temazepam 15 mg orally at bedtime
  Arms: temazepam
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to test two study drugs, one of which is temazepam (15mg) and one of which is a placebo (an inactive substance that looks just like the temazepam), to see if insomnia (trouble sleeping) can be reduced in patients with HIV infection. Placebos are given in research studies to try and make sure that subjects are responding to the effects of the study drug and not to other factors, like the attention they are receiving. If you decide to take part in this study, you will take 1 capsule of study drug every night approximately 30 minutes before bedtime for approximately 12 weeks.

This study is to test the study drug called temazepam for the treatment of insomnia (trouble sleeping) in patients with HIV infection. Temazepam has been approved by the FDA for the treatment of insomnia. However, because this study requires treatment for 12 weeks instead of the 7 to 10 days approved by the FDA, the use of temazepam is considered to be investigational in this study.

ELIGIBILITY:
Inclusion Criteria:

1. males or females age 18-69;
2. females must utilize an approved form of birth control during the study;
3. have at least a 3 month history of insomnia as defined in the DSM-IV criteria for primary insomnia;
4. self report > 60 minutes of wakefulness after initial sleep onset on at least 4 nights of 7 consecutive nights;
5. self report > 30 minutes of self-reported latency to sleep onset on at least 4 nights of 7 consecutive nights;
6. Self report < 6.5 hours of total sleep time at least 4 nights of 7 consecutive nights;
7. be able to read, understand, and sign an informed consent form before entering into the study and must be willing to comply with all study procedures;
8. agree to participate for the entire study period (a total of approximately 6 months); and
9. provide documentation of HIV seropositivity and be enrolled in ongoing care for their HIV disease in an infectious disease clinic with their last examination not exceeding 3 months prior to screening date

Exclusion Criteria:

1. Have a clinically significant unstable medical abnormality, or history or presence of significant neurological disorders (including cognitive disorders), or frequent nightly urination, defined as > 2 times per night;
2. Had a clinically significant illness, as determined by the Investigator, within 30 days of Initial Screening (Visit 1);
3. Have any clinically significant abnormal finding in physical examination, neurological assessment, or vital signs, as determined by the Investigator;
4. Have a known or exaggerated pharmacological sensitivity or hypersensitivity or intolerance to doxepin HCl, any tricyclic antidepressant or antihistamine, temazepam or any benzodiazepine;
5. Have a positive urine drug screen for amphetamines, benzodiazepines, barbiturates, cocaine, opiates, or cannabinoids at Initial Screening (Visit 1);
6. Self reports typical consumption of more than five alcoholic beverages on a single day or greater than 14 alcoholic beverages weekly;
7. Have a history of epilepsy or serious head injury;
8. Have been on current HAART or antiretroviral regimen for less than 1 month;
9. Have a recent history (within one year) of alcohol or drug abuse, or current evidence of substance dependence or abuse as defined by DSM-IV-TR criteria;
10. Have used temazepam for any indication within the 30 days prior to Initial Screening (Visit 1);
11. Have used any investigational drug within 30 days or five half-lives (whichever is longer) prior to Initial Screening (Visit 1), or plans to use an investigational drug (other than the study drug) during the study;
12. Current use of any of the following medications: antipsychotics, appetite suppressants, systemic corticosteroids, theophylline, respiratory stimulants and decongestants;
13. The following medications may be discontinued for the purpose of entry into the study provided the medication is taken at bedtime for the indication of sleep. If the indication is other than sleep, the medication cannot be discontinued for the purpose of entry into the study: anxiolytics, antidepressants, anticonvulsants, histamine-1 receptor antagonists (except for loratadine, desloratidine, and fexofenadine), narcotic analgesics, sedative/hypnotics (other than study drug) or OTC sleep aids;
14. Have symptoms consistent with the diagnosis of any other sleep disorder other than primary insomnia (e.g., sleep apnea, narcolepsy, periodic leg movements, restless leg syndrome, etc.);
15. Have a body mass index (BMI) greater than or equal to 34;
16. Have insomnia associated with circadian rhythm disturbances, such as night or rotating shift work or travel across more than four time zones in the 14 days before Initial Screening (Visit 1) or during the study;
17. Self reports intentional napping more than two times per week;
18. Have a variation in bedtime of more than three hours on five of seven consecutive nights as recorded on the sleep diary;
19. Have a history of non-adherence to treatment or clinical visit attendance; or,
20. subjects taking any benzodiazepine within 5 half-lives prior to the study baseline

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Krystal, MD, Principal Investigator — Duke University

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: After screening, all subjects meeting entry criteria will be placed on the same single blind study drug treatment, asked to complete a daily sleep diary, and return one week later. After one week subjects randomized to placebo will be given placebo for 12 weeks.
  Placebo
Period: Overall Study
Arm/Group | Temazepam | Placebo
Started | 25 | 19
Completed | 23 | 18
Not Completed | 2 | 1
Not completed — Physician Decision | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Temazepam | Placebo | Total
Number analyzed (Participants) | 25 | 19 | 44
Age, Customized [Number; unit: participants]
  21 - 69 years old | 25 | 19 | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 17 | 10 | 27
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 21 | 14 | 35
  Caucasian | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 25 | 19 | 44

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in the Insomnia Severity Index
Description: Mean change in the total score of the Insomnia Severity Index from Randomization to Final Study Visit after 12 weeks of double blind, placebo controlled dosing. The Insomnia Severity Index (ISI), is a 7-item questionnaire on a Likhert scale (0-4) assessing sleep initiation, sleep maintenance, satisfaction/distress over sleep problems, and daytime dysfunction. Responses to each item are summed to obtain a total score to determine the severity of insomnia. The total score can range from 0 to 28 with higher scores indicating greater insomnia severity.
Time Frame: Randomization to final study visit, approximately 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Temazepam | Placebo
Number analyzed (Participants) | 23 | 18
units on a scale | -4.01 (5.3) | 0.72 (6.1)

2. Secondary Outcome: Mean Change in Self Reported Total Sleep Time
Description: Mean change in self reported Total Sleep Time from Randomization to Final Study Visit in the placebo-controlled phase.
Time Frame: Randomization to final study visit, approximately 12 weeks
Population: Data not collected, and therefore not analyzed.
Arm/Group | Temazepam | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Mean Change in Self-reported Total Sleep Time
Description: Mean change in self-reported total sleep time from randomization to the end of the open label phase
Time Frame: Randomization to the end of the open label phase, approximately 1 week
Population: Data not collected, and therefore not analyzed.
Arm/Group | Temazepam | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Mean Change in Piper Fatigue Score
Description: A multidimensional scale for measuring fatigue, whose validity and reliability have been established across many patient populations including cancer patients, HIV, pregnancy, and myocardial infarction. There are 22 questions, in 3 subscales that measure behavioral, affective meaning, sensory and cognitive/mood aspects of fatigue, each scored on an 11-point likhert scale with a score of 0-10, 0 indicating no fatigue and 10 indicating the most severe fatigue. The Piper Fatigue Scale can range from 0 to 220 with higher scores indicating greater fatigue.
Time Frame: Baseline, week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Temazepam | Placebo
Number analyzed (Participants) | 23 | 18
units on a scale
  Baseline | 108 (48) | 126 (42)
  Week 12 | 57.9 (41) | 113 (46)

5. Secondary Outcome: Mean Change in the Hospital Anxiety and Depression Scale - Anxiety (HADS-A)
Description: A scale designed to detect states of anxiety and depression in the setting of an outpatient clinic, that consists of 2 sets: the HADS-A (Anxiety) and HADS-D (Depression). This is a series of 7 questions in each set (for a total of 14), assessed on a scale from 0-4, 0 being the response that indicates the least anxiety or depression, and 4 the most. Separate scores are calculated for anxiety and depression and a score (ranging from 0 to 21) is obtained for each subscale. The higher the score, the more severe the anxiety or depression.
Time Frame: Baseline, week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Temazepam | Placebo
Number analyzed (Participants) | 23 | 18
units on a scale
  Baseline | 7.1 (4.1) | 8.6 (4.0)
  Week 12 | 7.3 (5.3) | 7.1 (5.2)

6. Secondary Outcome: Mean Change in the Distress Thermometer
Description: A clinical tool that has been validated widely especially in cancer patients, to detect clinically significant emotional distress. This is a one-item scale that asks participants to rate their distress on scale from 0-100. Lower scores represent less distress and higher scores indicate greater distress.
Time Frame: Baseline, week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Temazepam | Placebo
Number analyzed (Participants) | 23 | 18
units on a scale
  Baseline | 44 (24.4) | 49.9 (25.3)
  Week 12 | 43 (26) | 39 (27)

7. Secondary Outcome: Mean Change in the Hospital Anxiety and Depression Scale - Depression (HADS-D)
Description: as for outcome 5
Time Frame: Baseline, week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Temazepam | Placebo
Number analyzed (Participants) | 23 | 18
units on a scale
  Baseline | 8.1 (4.2) | 8.1 (4.0)
  Week 12 | 7.3 (5.3) | 7.1 (5.2)

ADVERSE EVENTS:
Arm/Group | Temazepam | Placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/18
Other Adverse Events (participants affected / at risk) | 4/23 | 2/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Temazepam (N=23) | Placebo (N=18)
dry mouth (Gastrointestinal disorders) | 3 | 1
lethargy (Nervous system disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes